CLINICAL TRIAL: NCT05397535
Title: Traditional Exercise as Convenient Approach to Improve Health 1-Baduanjin Lower Elevated Blood PreSsure Study
Brief Title: Baduanjin Lower Elevated Blood PreSsure Study
Acronym: BLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-1724
Record Dates: First submitted 2022-05-20; First posted 2022-05-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Elevated Blood Pressure
Keywords: Baduanjin; elevated blood pressure; antihypertensive effect; randomized controlled trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Self-directed exercise group (No Intervention): Participants in the self-directed exercise group will choose the type and duration of exercise by their preference.
- Brisk walking group (Active Comparator): Participants in Brisk Walking Group will participate in brisk walking for 52 weeks (≥5 days/week, about 30 minutes/day).
  Interventions: Behavioral: Brisk walking
- Baduanjin group (Experimental): Participants in Baduanjin Group will practice Baduanjin singly for 52 weeks (≥5 days/week, about 30 minutes/day).
  Interventions: Behavioral: Baduanjin

INTERVENTIONS:
Behavioral: Baduanjin — Participants in Baduanjin group will receive health education on hypertension and attend a 4-hour class to learn Baduanjin before receiving the interventions after the randomization. Baduanjin exercise protocol is based on the "Fitness Qigong Baduanjin Standard" enacted by the General Administration of Sports in 2003. Each Badaunjin exercise session will last at least 30 minutes and be conducted at least 5 days per week for 52 weeks. These participants will be required to practice Baduanjin regularly, and the researchers will monitor their adherence to practice and provide reminders if needed.
  Arms: Baduanjin group
Behavioral: Brisk walking — Participants in this group will receive health education on hypertension and practice brisk walking on their own for at least 30 minutes, at least 5 days per week for 52 weeks. These participants will be required to do brisk walking regularly, and the researcher will monitor their adherence to practice and provide reminders if needed.
  Arms: Brisk walking group

SUMMARY:
The aim of this study is to evaluate the effects of Baduanjin on blood pressure in individuals with high normal blood pressure (SBP 130-139 mmHg, and/or DBP 85-89 mmHg), as well as on glucose and lipid metabolism, quality of life, psychology, exercise, immune inflammation, endothelial function, and arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older;
* Systolic blood pressure (SBP) <140 mmHg and diastolic blood pressure (DBP) <90 mmHg
* SBP 130-139 mmHg, and/or DBP 85-89 mmHg

Exclusion Criteria:

* Diagnosis of hypertension (SBP≥140 mmHg, and/or DBP ≥90mmHg）
* History of cardiovascular diseases, such as coronary heart disease, heart failure, stroke, and peripheral vascular disease
* Diagnosis of chronic kidney disease, primary aldosteronism, Cushing's syndrome, or pheochromocytoma
* Newly diagnosed cancer or cancer metastasis within 5 years
* History of autoimmune disease
* Having taken antihypertensive drugs or immunoregulators within 2 weeks
* A long-term need for antihypertensive drugs or immunomoregulators
* Unable to maintain moderate intensity exercise due to illness or other reasons
* Pregnant, breastfeeding, or planning to become pregnant within the next 1 year
* Currently taking regular exercise (at least 30 minutes of moderate-intensity exercise at least three times a week)
* Allergic to sports bracelets
* Having participated or been participating in other clinical trials within the last 3 months
* Unable to use smartphones
* Other factors that may affect the follow-up, such as alcohol or substance abuse in the last 12 months, planing to live out of town for a long time, or diagnosis of dementia or cognitive impairment which indicates incapability of completing the study
* Unable to accurately measure blood pressure using the sphygmomanometer provided by the study due to a too large or too small arm circumference

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline ambulatory 24-h systolic blood pressure (mmHg) at 12 week | Baseline, 12 week
  Change form Baseline ambulatory 24-h systolic blood pressure at 12 week will be measured by ambulatory blood pressure monitoring to investigate the short-term antihypertensive effect of Baduanjin.
Change from baseline ambulatory 24-h systolic blood pressure (mmHg) at 52 week | Baseline, 52 week
  Change from baseline ambulatory 24-h systolic blood pressure at 52 week will be measured by ambulatory blood pressure monitoring to investigate the long-term antihypertensive effect of Baduanjin.

SECONDARY OUTCOMES:
Other blood pressure indicators: daytime mean SBP(mmHg), nighttime mean SBP(mmHg), 24-h DBP(mmHg), daytime mean DBP(mmHg), nighttime mean DBP(mmHg) | Baseline,12 week,52 week
  Other blood pressure indicators:daytime mean systolic blood pressure, nighttime mean systolic blood pressure, 24-h diastolic blood pressure, daytime mean diastolic blood pressure, nighttime mean diastolic blood pressure
SBP(mmHg) | Baseline,4 week,8 week,12 weeks,24 week,32 week,52 week
  Blood pressure indicator:office systolic blood pressure
DBP(mmHg） | Baseline,4 week,8 week,12 weeks,24 week,32 week,52 week
  Blood pressure indicator:office diastolic blood pressure
FBG(mmol/L) | Baseline,12 week,52 week
  Glucose metabolism indicator: fasting blood glucose
HbA1c(%) | Baseline,12 week,52 week
  Glucose metabolism indicator: hemoglobin A1c
Insulin | Baseline,12 week,52 week
  Glucose metabolism indicator
C-peptide | Baseline,12 week,52 week
  Glucose metabolism indicator
Lipid metabolism parameters: TC(mmol/L), TG(mmol/L), HDL-C(mmol/L), LDL-C(mmol/L) | Baseline,12 week,52 week
  Lipid metabolism indicators: total cholesterol , triglyceride , high density lipoprotein cholesterol, low density lipoprotein cholesterol
Total scores of The Short-Form-36 Health Survey (SF-36) | Baseline,12 week,52 week
  The total scores range from 0-100, and the higher scores mean better outcomes
Total scores of Pittsburgh Sleep Quality Index(PSQI) | Baseline,12 week,52 week
  The total scores range from 0-21, and the higher scores mean worse outcomes
Total scores of Generalized Anxiety Disorder-7(GAD-7) | Baseline,12 week,52 week
  The total scores range from 0-21, and the higher scores mean worse outcomes
Total scores of Patient Health Questionnaire-9 items(PHQ-9) | Baseline,12 week,52 week
  The total scores range from 0-27 , and the higher scores mean worse outcomes
Total scores of Neck Disability Index(NDI) | Baseline,12 week,52 week
  The total scores range from 0-100%, and the higher scores mean worse outcomes
Sit and reach test(cm) | Baseline,12 week,52 week
  Motor system function: sit and reach test

OTHER OUTCOMES:
hs-CRP(mg/L) | Baseline,12 week,52 week
  Inflammatory indicator:high-sensitivity C-reactive protein
IL-1β(pg/mL) | Baseline,12 week,52 week
  Inflammatory indicator:interleukin-1β
TNF-α(pg/mL) | Baseline,12 week,52 week
  Inflammatory indicator:tumor necrosis factor-α
FMD(%) | Baseline,12 week,52 week
  Endothelial function indicator:flow mediated dilatation
NO(μmol/mL) | Baseline,12 week,52 week
  Endothelial function indicator:nitric oxides
PG(pg/mL) | Baseline,12 week,52 week
  Endothelial function indicator:prostaglandin
cfPWV(m/s) | Baseline,12 week,52 week
  Atherosclerosis:carotid-femoral pulse wave velocity
Whole genome gene expression profiling in peripheral blood mononuclear cells | Baseline,12 week,52 week
  Immunological indicator
Thymic volume(cm^3) | Baseline,52 week
  Immunological indicator
BMI(kg/m^2) | Baseline,12 week,52 week
  Anthropometric indicator:Body mass index
Waist circumference(cm) | Baseline,12 week,52 week
  Anthropometric indicator

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD,PhD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No